CLINICAL TRIAL: NCT01828593
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Clinical Study Evaluating the Impact of Serum-derived Bovine Immunoglobulin Protein Isolate, a Medical Food, on Nutritional Status in HIV+ Subjects With HIV-associated Enteropathy.
Brief Title: Impact of SBI, a Medical Food, on Nutritional Status in Patients With HIV-associated Enteropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entera Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EH6001
Record Dates: First submitted 2013-04-08; First posted 2013-04-10 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-04

CONDITIONS: HIV-associated Enteropathy
MeSH Terms: conditions — HIV Enteropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Other: Placebo
- SBI 2.5 g (Active Comparator): Serum-derived bovine immunoglobulin protein isolate (SBI) 2.5 g
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
- SBI 5.0g (Active Comparator): Serum-derived bovine immunoglobulin protein isolate (SBI)5.0g
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin protein isolate (SBI) — SBI is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
  Arms: SBI 2.5 g; SBI 5.0g
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the oral nutritional therapy serum-derived bovine immunoglobulin protein isolate (SBI) 2.5 g twice a day (BID) and SBI 5.0 g versus placebo on supporting nutrient absorption in HIV+ subjects with HIV-associated enteropathy.

DETAILED DESCRIPTION:
This study is evaluating the effectiveness of the oral nutritional therapy serum-derived bovine immunoglobulin protein isolate (SBI) 2.5g BID and SBI 5.0g compared to placebo for 6 months on gastrointestinal symptoms, nutritional status and quality of life in HIV+ subjects with HIV-associated enteropathy. In addition, the effects of SBI on pro-inflammatory intestinal microbial populations, bacterial translocation, intestinal barrier function, and systemic immune activation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* History of HIV-1 infection
* Plasma HIV viral load ≤40 copies/mL
* Maintained virologic suppression for 1 year
* Stable Antiretroviral Therapy (ART) regimen
* History of HIV-associated diarrhea defined as abnormal passage of 3 or more unformed stools per day or a liquid stool volume greater than 200 g per day for at least 4 weeks duration

Exclusion Criteria:

* Positive stool test for pathogenic bacteria, C. difficile or ova and parasites
* Conditions that require chronic therapy that is known to alter gut microbiota
* Antibiotics within 2 weeks of screening (exception: prophylaxis antibiotics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Asmuth, M.D., Principal Investigator — University of California, Davis
Locations (10):
- United States (10):
  - AIDS Research Alliance, Los Angeles, California
  - Univ of California Davis CARES Clinic, Sacramento, California
  - Univ of California SF, San Francisco, California
  - Therafirst, Fort Lauderdale, Florida
  - Miami Springs, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - Cincinnati, Ohio
  - Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consists of 2 phases, the Placebo-controlled (PC) phase and the Placebo-free (PF) extension phase. Participants were randomized in a 1:1:2:2 ratio into 4 groups: Placebo for 4 wk PC phase followed by either 2.5g or 5.0g BID for 20 wk PF phase or SBI 2.5g or 5.0g BID for 4-wk PC phase followed by 2.5g or 5.0g for 20 wk PF phase.
Groups:
- Placebo: Matching Placebo
  Following 4 weeks in placebo-controlled phase were randomized to either SBI 2.5 g or SBI 5.0 g
Period: Placebo-Controlled Phase
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0g
Started | 36 | 34 | 33
Completed | 36 | 34 | 32
Not Completed | 0 | 0 | 1
Period: Placebo-Free Phase
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0g
Started | 0 (Placebo subjects took either SBI 2.5 or 5.0 g in the placebo-free phase) | 55 (SBI 2.5 g includes SBI 2.5 plus placebo who started taking SBI at Wk 4) | 47 (SBI 5.0 g includes SBI 5.0 plus placebo who started taking SBI at Wk 4)
Completed | 0 (Placebo subjects took either SBI 2.5 or 5.0 g in the placebo-free phase) | 49 (SBI 2.5 g includes SBI 2.5 plus placebo who started taking SBI at Wk 4) | 41 (SBI 5.0 g includes SBI 5.0 plus placebo who started taking SBI at Wk 4)
Not Completed | 0 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0g | Total
Number analyzed (Participants) | 36 | 34 | 33 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (6.8) | 50.9 (6.7) | 50.7 (8) | 51.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 11 | 32
  Male | 28 | 21 | 22 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 11
  Not Hispanic or Latino | 32 | 29 | 31 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 20 | 22 | 63
  White | 14 | 14 | 10 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Years with HIV [Mean (Standard Deviation); unit: years] | 16 (7.6) | 16.9 (6.3) | 17.9 (6.3) | 16.9 (6.76)
Years with HIV-associated diarrhea [Mean (Standard Deviation); unit: years] | 4.4 (5.4) | 6.9 (7.3) | 6.6 (6.7) | 5.9 (6.54)
Baseline Plasma CD4+ cell count [Mean (Standard Deviation); unit: cells/microliter] | 629 (307) | 746 (324) | 671 (319) | 682 (317)
Plasma viral load [Mean (Standard Deviation); unit: copies/mL] | 24 (11) | 27 (22) | 28 (28) | 26 (21)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Daily Unformed Bowel Movements
Description: Change in number of abnormal or unformed stools by week 4
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: abnormal or unformed stools
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0g
Number analyzed (Participants) | 36 | 34 | 33
abnormal or unformed stools | -2.46 (2.01) | -2.16 (2.18) | -2.20 (1.99)

2. Other Pre Specified Outcome: Change From Baseline in Peripheral CD4+ T Cell Counts in Lowest Baseline CD4+ Quartile (Less Than or Equal to 418)
Description: Lowest baseline CD4+ quartile (less than or equal to 418)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cells/microliter
Groups:
- SBI 2.5 g: Serum-derived bovine immunoglobulin protein isolate (SBI) 2.5 grams
  Serum-derived bovine immunoglobulin protein isolate (SBI): SBI is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
- SBI 5.0 g: Serum-derived bovine immunoglobulin protein isolate (SBI) 5.0 grams
  Serum-derived bovine immunoglobulin protein isolate (SBI): SBI is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0 g
Number analyzed (Participants) | 10 | 7 | 8
cells/microliter | -19.8 (59.22) | 41.86 (84.83) | 47.63 (42.63)

3. Other Pre Specified Outcome: Change From Baseline in Peripheral CD4+ T Cell Counts in 2nd Baseline CD4+ Quartile (Greater Than 418 and Less Than or Equal to 630
Description: 2nd Baseline CD4+ Quartile (greater than 418 and less than or equal to 630)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0 g
Number analyzed (Participants) | 13 | 6 | 6
cells/microliter | 31.46 (122.70) | 82.67 (205.16) | 12.00 (119.75)

4. Other Pre Specified Outcome: Change From Baseline in Peripheral CD4+ T Cell Counts in 3rd Baseline CD4+ Quartile (Greater Than 630 and Less Than or Equal to 890)
Description: 3rd Baseline CD4+ Quartile (Greater than 630 and Less than or Equal to 893)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0 g
Number analyzed (Participants) | 1 | 10 | 13
cells/microliter | 48.00 (NA) | 36.70 (183.14) | -29.46 (224.83)

5. Other Pre Specified Outcome: Change From Baseline in Peripheral CD4+ T Cell Counts in 4th Baseline CD4+ Quartile (Greater Than 893)
Description: 4th Baseline CD4+ Quartile (greater than 893)
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | Placebo | SBI 2.5 g | SBI 5.0 g
Number analyzed (Participants) | 10 | 10 | 4
cells/microliter | -144.00 (155.15) | -54.20 (230.43) | -365.25 (464.04)

6. Other Pre Specified Outcome: Change From Baseline in Duodenal Gut-associated Lymphoid Tissue (GALT) CD4+ T Cell Densities
Time Frame: Baseline and Week 24
Population: Sub-study
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | CD4 + T Cell Counts | CD8 + T Cell Counts
Number analyzed (Participants) | 8 | 8
cells/mm3 | 144.80 [-107.5 to 324.7] | -67.95 [-339.4 to 187.9]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- SBI 2.5 g: Serum-derived bovine immunoglobulin protein isolate (SBI) 2.5 g - Subjects on 2.5 g in the placebo controlled phase and placebo free phase and subjects who went from placebo in the placebo controlled phase to 2.5 g in the placebo free phase
  Serum-derived bovine immunoglobulin protein isolate (SBI): SBI is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
- SBI 5.0g: Serum-derived bovine immunoglobulin protein isolate (SBI)5.0g - Subjects on 5.0 g in the placebo controlled phase and placebo free phase and subjects who went from placebo in the placebo controlled phase to 5.0 g in the placebo free phase
  Serum-derived bovine immunoglobulin protein isolate (SBI): SBI is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. SBI does not contain any milk products such as lactose, casein, or whey. SBI is gluten-free, dye-free, and soy-free. SBI is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
Arm/Group | SBI 2.5 g | SBI 5.0g
Serious Adverse Events (participants affected / at risk) | 2/55 | 1/47
Other Adverse Events (participants affected / at risk) | 26/55 | 20/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBI 2.5 g (N=55) | SBI 5.0g (N=47)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBI 2.5 g (N=55) | SBI 5.0g (N=47)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (General disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Blood Glucose Increased (Investigations) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no multi-site publication is made within 18 months, Site may publish Site's results, subject to the following. At least 30 days prior to submitting a manuscript the Site shall provide to Entera a copy, and Entera shall have 30 days to review. Site shall remove any Confidential Information, upon Entera's request, prior to submitting the materials, and the Site shall delay publication for an additional period of up to 60 days to allow Entera to protect its interests in any Inventions.